CLINICAL TRIAL: NCT04216745
Title: Microbial Profile of Cholangitis in Patients Undergoing Biliary Intervention
Brief Title: Microbial Analysis in Patients With Cholangitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nourhan Mostafa Salama, Assistant Lecturer, Assiut University
Other Study IDs: Microbial profile in bile
Record Dates: First submitted 2019-12-27; First posted 2020-01-03 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Cholangitis
MeSH Terms: conditions — Cholangitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: bile culture — Bile samples will be collected for microbial cultures and antimicrobial susceptibility testing using COMPACT-15 automated system (Bio Merieux, Marcy I'Etoile, France) for bacteria and saboroud's agar for fungal culture.

SUMMARY:
* To identify the microbial profile in bile and blood for patients with cholangitis.
* To explore risk factors of cholangitis and outcomes in those patients

DETAILED DESCRIPTION:
Under physiological conditions, bile is sterile. Major factors maintaining sterility of bile are a competent sphincter of Oddi and antegrade flow of bile. Other factors are bile salts in the bile duct, Kupffer cells and tight junctions between the hepatocytes that guard against bacteria getting in from the portal circulation. Any break in these physiological barriers leads to infection of the bile. The main source of infection in most cases is the duodenum. Hematogenous spread through the portal venous flow is another route. In addition, bile duct obstruction e.g., stone, is associated with bacterial colonization within the stagnant bile and with increasing biliary pressure, bacteria may translocate into the circulation causing a systemic infection .

In patients without stone disease, previous biliary intervention is associated with high rates of infection. Bacteremia as a complication of biliary intervention tends to occur in patients with obstructed bile flow, especially those who have previously undergone orthotopic liver transplantation (OLT), surgery to the biliary tree, sphincterotomy, or placement of a biliary stent. The risk of systemic infection is high when adequate biliary drainage has not been achieved after intervention, which typically involves endoscopic retrograde cholangiopancreatography (ERCP) or percutaneous transhepatic cholangiography (PTC).

Acute cholangitis is acute inflammation and infection in the bile duct. It is diagnosed in 6-9% of patients with gallstone disease and 1-3% after ERCP. It can progress from a local biliary infection to advanced systemic disease with sepsis and multiple organ dysfunctions with significant mortality rates (10%).

Microbial infection causing acute cholangitis is mainly bacteria and fungi. Despite blood cultures provide an opportunity to detect the causative organism, they remain negative in more than half of the cases with cholangitis. The growth is often mono-microbial organism, predominantly Gram-negative organisms. However, bile cultures often have a poly-microbial growth especially in patients with an indwelling biliary stent where, Gram-negative bacteria, in particular Escherichia coli, are the most common pathogens isolated from infected bile.

The fungal infection of the biliary tract increase in the last years and can lead to biliary obstruction. The most common fungal infection in biliary tract is candidiasis.

Because of the rapid development of multi-drug resistant organisms, the choice of appropriate empiric antimicrobial therapy has become more complicated. Thus, knowledge of the common etiologic agents and their local susceptibility profile is essential to ensure the appropriate choice and timely administration of empiric antimicrobial therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with extrahepatic cholestasis undergoing biliary procedure (ERCP or PTD) will be included.

Exclusion Criteria:

* patients less than 18 years old.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - Patients with extrahepatic cholestasis undergoing biliary procedure (ERCP or PTD)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the microbial profile of cholangitis | Up to 24 weeks
  to evaluate the microbial profile of cholangitis regarding types of organisms

SECONDARY OUTCOMES:
Evaluation of short-term mortality | Up to 24 weeks
  follow up patients with cholangitis to evaluate short-term mortality rate (%)

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Sharaf, AP, Study Director — Assiut University
Locations (1):
- Assiut, Asyut, Egypt